CLINICAL TRIAL: NCT01679795
Title: Vascular Effect of Tibolone Versus Placebo Evaluated by Flow-mediated Dilatation of Brachial Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, Associate Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDILA
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Flow-mediated Dilation Evaluation of the Brachial Artery
Keywords: hormone replacement therapy; Dopplervelocimetry; Flow-mediated dilation; menopause; tibolone
MeSH Terms: interventions — tibolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Tibolone (Experimental): patientes will use tibolone 2,5mg/day during 30 days
  Interventions: Drug: Tibolone
- Placebo use (Placebo Comparator): Patients will use placebo for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tibolone
  Other Names: Livial
  Arms: Tibolone
Drug: Placebo
  Arms: Placebo use

SUMMARY:
The aim of this study is to evaluate the vascular effects of tibolone on climateric women measured by flow-mediated evaluation of the brachial artery using high resolution ultrasound and compare to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women without menstrual cycles whithin the last 12 months and FSH>30IU/L
* Healthy women
* Women that were not using drugs with potential vascular effect whithin the last 1 year
* Women that never used hormone replacement therapy

Exclusion Criteria:

* Smoking
* Blood Pressure > 160/90 mm Hg.
* Breast and or endometrial cancer
* History of acute myocardial infarction
* Diabetes
* Vaginal bleeding of any origin
* Hepatic disease
* thrombophlebitis or thromboembolic disorders

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the brachial artery one month after treatment started Flow-mediated dilation of the brachial artery one month after treatment started Flow-mediated dilation of the brachial artery | 30 days
  Flow-mediated dilation will be measured by high resolution ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil